CLINICAL TRIAL: NCT00262548
Title: Interventions Study for the Control of Diabetes Mellitus Type 2 in Obese Women
Brief Title: C-Reactive Protein (CRP) in Obese Diabetic Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Mexican National Institute of Public Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DM-CRESTOR-0001; D3560L00018
Record Dates: First submitted 2005-10-26; First posted 2005-12-07 (Estimated); Last update posted 2007-08-28 (Estimated); Status verified 2007-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Obesity; Menopause
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — Rosuvastatin Calcium

INTERVENTIONS:
Drug: Rosuvastatin; improvement of lipid profile

SUMMARY:
The purpose of this study is to determine whether treatment with rosuvastatin for 6 months in obese type 2 diabetic women will improve their lipid profiles and thus prevent the progression to cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Menopausal
* Diagnosed diabetes mellitus type 2
* Obese (body mass index [BMI] > 25 ≤ 30)

Exclusion Criteria:

* Fasting blood glucose ≥ 200 mg/dl
* CRP < 2 mg/L and > 10 mg/L

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-10

PRIMARY OUTCOMES:
Patients will be receiving rosuvastatin/placebo for 6 months
They will have baseline laboratory parameters taken such as glycemia
HbA1c (glycosylated hemoglobin), low-density lipoprotein cholesterol (LDL-C), computed tomography (CT), high-density lipoprotein cholesterol (HDL-C), C-reactive protein (CRP), and retaken every 3 months
Every month, patients will be evaluated at the clinic
All participants will receive an intervention on diet and physical activity counseling, which will be carefully monitored.

SECONDARY OUTCOMES:
Other variables will be: proinflammatory cytokines - tumor necrosis factor (TNF)-alpha, interleukin-6 (IL-6), IL-12, Th2/Th3 cytokines -IL-4, IL-10 and transforming growth factor beta (TGF-beta)

CONTACTS AND LOCATIONS:
Overall Officials: Astra Zeneca Mexico Medical Director, MD, Study Director — AstraZeneca; Simón Barquera Cervera, MD, Principal Investigator — Mexican National Institute of Public Health
Locations (1):
- Research site, Cuernavaca, Morelos, Mexico